CLINICAL TRIAL: NCT03723694
Title: Dietary Modulation of Neuroinflammation in Age-Related Memory Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Richard P Sloan PhD, Nathaniel Wharton Professor of Behavioral Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NYSPI 7665; 5R01AG058417 (NIH)
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Memory Loss; Inflammation
Keywords: Flavanol; Cocoapro
MeSH Terms: conditions — Memory Disorders; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 650 mg of Cocoapro flavanols (Active Comparator): Daily, each subject will consume either two cocoa flavanol-containing capsules twice a day with a meal.
  Interventions: Dietary Supplement: 650 mg of Cocoapro flavanols
- 0mg Cocoapro flavanols (Placebo Comparator): Daily, each subject will consume either ttwo placebo-containing capsules twice a day with a meal.
  Interventions: Dietary Supplement: 0 mg of Cocoapro flavanols

INTERVENTIONS:
Dietary Supplement: 650 mg of Cocoapro flavanols — 12-week period during which participant will be asked to consume two cocoa-flavanol-containing capsules(650mg) twice a day with meals.
  Arms: 650 mg of Cocoapro flavanols
Dietary Supplement: 0 mg of Cocoapro flavanols — 12-week period during which participant will be asked to consume two cocoa-flavanol-containing capsules(0mg) twice a day with meals.
  Arms: 0mg Cocoapro flavanols

SUMMARY:
The purpose of this study is to test the effect of a cocoa-derived dietary flavanol on brain structures and cognitive outcomes in a 12-week randomized controlled trial of 146 healthy participants, age 50-69, who will receive this cocoa derivative or a placebo. Th investigators will also examine the role of inflammation in this relationship.

DETAILED DESCRIPTION:
Within 25 years, the US population aged 65 and over will double in size to 80 million bringing, with it an epidemic of aging-related cognitive decline, from normal cognitive aging to neurodegenerative disorders including Alzheimer's Disease. These conditions impair quality of life and functional status, impose an enormous burden on individuals, their families, the healthcare system, and require elucidation of mechanisms and development of new treatments to prevent or at least slow their progression. The use of plant-based food and drink for health purposes has a long and well-documented history. Cocoa beans contain a substance that has multiple beneficial health effects. In this study, the investigators will test the effect of this substance on brain structures and cognitive outcomes in a 12-week randomized controlled trial of 146 healthy participants, age 50-69, who will receive this cocoa derivative or a placebo. The investigators also will examine the role of inflammation in this relationship. Such a trial has potential for significant clinical impact.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal screening or management of the subject).
2. Healthy Male or Female subjects. (Females must be post-menopausal)
3. Age between 50 and 69 years, both inclusive.
4. Body mass index between 18.0 and 35 kg/m², both inclusive.

Exclusion Criteria:

1. Currently undergoing medical treatment, including prescription drugs/medication.
2. Clinically significant abnormal hematology, biochemistry, urinalysis, or coagulation screening tests, as judged by the Investigator.
3. History or presence of cancer (except basal cell skin cancer or squamous cell skin cancer), or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological (with the exception euthyroid struma), haematological, dermatological, venereal, neurological, psychiatric diseases or other major disorders as judged by the Investigator.
4. Seated blood pressure at screening (after resting for 5 min in seated position) outside the range of 90-140 mmHg for systolic or 50-90 mmHg for diastolic (excluding white-coat hypertension; therefore, if a repeated measurement shows values within the range, the subject can be included in the trial) and/or resting supine heart rate outside the range 50-90 beats per minute. Measurement taken at consent before eligibility is determined
5. Heart Diseases.
6. Hepatitis B or C positive status.
7. HIV positive status.
8. History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
9. Use of non-prescription medication, herbal products or nutritional supplements during the study, and within the last 4 weeks before the start of the study (screening), as judged by the Investigator; occasional use of aspirin, ibuprofen, acetaminophen is permitted.
10. Adherence to a vegan or vegetarian diet or to specialty/uncommon diets.
11. Food Allergies to tree nuts, soy, cocoa and cocoa-containing products.
12. People who choose to avoid caffeine intake.
13. Current or history of alcoholism or drug/chemical abuse as per Investigator's judgment.
14. Hormone Replacement Therapy; Currently pregnant; Pregnant or Interview\ lactating within past 6 months; Hormonal birth control (pill).
15. Smoking.
16. Unwilling to have blood drawn or anxiety/nausea during a blood draw.
17. Uncomfortable completing memory and attention tasks in the English language
18. Montreal Cognitive Assessment (MoCA) score less than 26.
19. Inability to swallow study capsules Interview (at Consent)
20. Did not complete the two weeks Run-In Period (Participants who missed more than 2 intake occasions out of 14 days (28 occasions total) or if there are > 8 capsules left in the bottle after the two weeks will be excluded).

MRI RELATED

1. Cardiac Pacemaker
2. Internal Pump
3. Insulin Pump
4. Tattoo eyeliner
5. Wire sutures
6. Internal Metal Objects
7. Metal Slivers in Eye
8. Prosthesis
9. Hearing Aid Implants
10. Neurostimulator
11. Metal Fragments
12. Brain Aneurysm Clips
13. Vascular Clips
14. Breast Expander
15. Vena Cava Filter
16. Heart Valve
17. Metal Stents
18. Asthmatic symptoms within the past 3 years
19. Sickle Cell Disease

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
HMGB1 | 12 weeks
  circulating levels of the inflammatory marker HMGB1

SECONDARY OUTCOMES:
NFkB | 12 weeks
  TLR4-dependent NFkB
TNFa | 12 weeks
  TLR4-dependent TNFa

OTHER OUTCOMES:
ModBent | 12 weeks
  modified Benton Recognition Task
ModRey | 12 weeks
  Modified Rey Auditory Verbal Learning Test
multiple cognitive domains | 12 weeks
  NIH Toolbox Cognition Battery, which includes adaptive computerized tests of executive function, attention, episodic memory, language, processing speed, and working memory

CONTACTS AND LOCATIONS:
Overall Officials: Richard P. Sloan, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

REFERENCES:
- [Background] Brickman AM, Khan UA, Provenzano FA, Yeung LK, Suzuki W, Schroeter H, Wall M, Sloan RP, Small SA. Enhancing dentate gyrus function with dietary flavanols improves cognition in older adults. Nat Neurosci. 2014 Dec;17(12):1798-803. doi: 10.1038/nn.3850. Epub 2014 Oct 26. PMID 25344629